CLINICAL TRIAL: NCT02210390
Title: Feasibility RCT of the Efficacy of a Culturally Adapted Psychological Intervention for Bipolar Disorder in Pakistan
Brief Title: Culturally Adapted Psychological Intervention for Bipolar Disorder in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other); Dow University of Health Sciences (Other); Abbasi Shaheed Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY-BPD-03
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Bipolar Disorder
Keywords: Psycho-education, Bipolar , cultural adaptation, Pakistan
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Psycho-education Sessions will be offered weekly basis
  Interventions: Behavioral: Psycho education
- Control (No Intervention): Patients who will be randomized to the "treatment as usual" arm will receive routine care

INTERVENTIONS:
Behavioral: Psycho education — Psycho-education Sessions will be offered weekly basis
  Arms: Intervention

SUMMARY:
Aim:

To assess the Feasibility RCT of the efficacy of a culturally adapted psychological intervention for Bipolar disorder in Pakistan

Design:

Randomized Control Trial

Setting:

Psychiatric Departments of different Hospitals in Karachi.

Participants:

A total of 36 Bipolar disorder patients will be randomized to psychological Intervention and treatment as usual arm.

Intervention:

Culturally Adapted psychological intervention for bipolar disorder

Outcome measure:

* Acceptance of intervention in terms of attending session and dropouts
* Knowledge and attitudes towards bipolar disorder

DETAILED DESCRIPTION:
The purpose of the study is to test Feasibility RCT of the efficacy of a culturally adapted psychological intervention for Bipolar disorder in Pakistan

Primary Objectives :

1. To determine effectiveness of educational intervention in terms of patient Satisfaction with overall care, knowledge and attitudes to bipolar disorder and medication adherence.
2. To assess feasibility in terms of

   * Recruitment
   * Using instruments that will be used to assess recurrence rate in the main study (BDI, YMRS and obtaining prospective hospitalisation and medication data)
   * acceptability of a culturally adapted bipolar group education package
3. To allow 'fine tuning' of culturally adapted bipolar group education package (this will partly be achieved by using the SEMI at study entry)

The Participants will be recruited from psychiatric department of different hospitals.

They will be randomly divided into two groups; intervention group and treatment-as-usual group. A total of thirty six participants will be recruited in the pilot study and divided equally into two arms. This will ensure that, even after loss to follow-up, we will have at least 12 subjects per group for analysis (FDA guidance http://www.fda.gov/cder/guidance/5356fnl.pdf) .Randomization will be carried out by the on offsite statistician. This will provide a reliable geographically remote service. For intervention group twelve sessions of psychoeducation will be provided by trained research clinician during the period of three months. Patients in the treatment as usual (TAU) group will be given details of intervention at the end of the study and interested patients will be offered psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM IV Bipolar disorder
* Currently stable (YMRS <8, BDI<12)
* Age 18 to 65 years.
* Participants engaged with the mental health services since last 6 months.
* Able to give written informed consent.
* Resident of trial catchments area
* Ability to speak Urdu /Punjabi

Exclusion Criteria:

* Substance or alcohol dependent (i.e., those who fulfill the criteria for dependence according to DSM IV criteria)
* Inability to engage fully in the psychotherapy (due to cognitive impairment)
* Actively suicidal
* Any major psychiatric illness other than bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale(YMRS) | three months
  The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms
Knowledge and attitudes | three months
  Knowledge and attitudes towards bipolar disorder measured by using a standard questionnaire
Beck's Depression Inventory Scale (BDI) | three months
  The BDI is a measure of depression severity and has been used in several previous studies in Pakistan and is validated for use in Urdu.

SECONDARY OUTCOMES:
Medication adherence | three months
  Self-reported Measure of Medication adherence
Visual Analogue Scale | three months
  Patient satisfaction with overall care
Short Explanatory Model Interview | three months
  used to elicit beliefs of mental illness

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, MD, Principal Investigator — Pakistan Institute of Learning and Living, University of Manchester; Imran Chaudhry, MD, Principal Investigator — University of Manchester; Farooq Naeem, MRCPsych, Principal Investigator — Pakistan Institute of Learning and Living, University of Southampton; Raza Ur Rehman, FCPS, Principal Investigator — Dow University of Health Sciences; Ajmal kazm, Principal Investigator — Pakistan Institute of Living and Learning; Munir Hamirani, FCPS, Principal Investigator — Abbasi Shaheed Hospital; Muhammad I Husain, MRCPsych, Principal Investigator — Camden and Islington NHS Foundation Trust
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Husain MI, Chaudhry IB, Rahman RR, Hamirani MM, Mehmood N, Haddad PM, Hodsoll J, Young AH, Naeem F, Husain N. Pilot study of a culturally adapted psychoeducation (CaPE) intervention for bipolar disorder in Pakistan. Int J Bipolar Disord. 2017 Dec;5(1):3. doi: 10.1186/s40345-017-0074-8. Epub 2017 Feb 11. PMID 28155203